CLINICAL TRIAL: NCT02315807
Title: Neurostimulation for Cognitive Enhancement After Stroke (NeuroCog)
Brief Title: Neurostimulation for Cognitive Rehabilitation in Stroke
Acronym: NeuroCog
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Suellen Marinho Andrade, PhD, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NeuroCog001
Record Dates: First submitted 2014-12-09; First posted 2014-12-12 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Stroke; Cognitive Impairment; Cerebral Infarction
MeSH Terms: conditions — Stroke; Cognitive Dysfunction; Cerebral Infarction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- dlPFC (Experimental): Participants in the chronic post-stroke stage will receive active transcranial direct current stimulation in dorsolateral prefrontal cortex
  Interventions: Device: transcranial direct current stimulation
- CON (Experimental): Participants in the chronic post-stroke stage will receive active transcranial direct current stimulation in cingulo-opercular network
  Interventions: Device: transcranial direct current stimulation
- M1 (Active Comparator): Participants in the chronic post-stroke stage will receive active transcranial direct current stimulation in motor primary cortex
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation
  Other Names: tdcs

SUMMARY:
Transcranial direct current stimulation has shown promising results in stroke patients. This study is a double blind, sham-controlled clinical trial aiming to compare the long-term effects of stimulation in two different cognitive regions after a stroke. Sixty patients who suffer from chronic strokes will be randomized into 1 of 3 groups: dorsolateral prefrontal cortex, cingulo-opercular network and motor primary cortex (control). Each group will receive transcranial direct current stimulation for 20 minutes for 10 consecutive working days (2 weeks). Patients will be assessed with a Dysexecutive Questionnaire, Semantic Fluency test, categorical verbal fluency and Go-no go tests, Wechsler Adult Intelligence Scale, Rey Auditory-Verbal Learning Test, Letter Comparison and Pattern Comparison Tasks at baseline, after their tenth stimulation session (week 2) and endpoint (week 4). Those who achieve clinical improvement with neurostimulation will be invited to receive treatment for 12 months as part of a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

* Ischaemic chronic stroke
* Mild/Moderate Cognitive impairment
* Informed consent

Exclusion Criteria:

* National Institute of Health Stroke Scale (NIHSS) ≥ 16 points
* Severe cognitive comorbidities (dementia, depression)
* transcranial direct current stimulation criteria: use of modulators of the Central Nervous System drugs; patients with implanted metallic or electronic devices; pacemaker; seizures; pregnancy;any other condition that might limit or interfere in the sensorimotor system

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Executive Function measured by Dysexecutive Questionnaire (DEX) | Change for executive functions at 4 weeks

SECONDARY OUTCOMES:
Verbal Fluency (Semantic Fluency Test) | [ Time Frame: Baseline, Week 2 and Week 4 ]
Response inhibition (Go-no-go Test) | [ Time Frame: Baseline, Week 2 and Week 4 ]
Executive function (Wechsler Intelligence Scale for Adults) | [ Time Frame: Baseline, Week 2 and Week 4 ]
Memory (Rey Auditory Verbal Learning) | [ Time Frame: Baseline, Week 2 and Week 4 ]
Processing Speed (Letter Comparison and Pattern Comparison Tasks) | [ Time Frame: Baseline, Week 2 and Week 4 ]

CONTACTS AND LOCATIONS:
Overall Officials: Suellen Andrade, PhD, Principal Investigator — Federal University of Paraíba
Locations (1):
- Suellen Andrade, João Pessoa, Paraíba, Brazil

REFERENCES:
- [Derived] Andrade SM, Fernandez-Calvo B, Boggio PS, de Oliveira EA, Gomes LF, Pinheiro Junior JE, Rodrigues RM, de Almeida NL, Moreira GM, Alves NT. Neurostimulation for cognitive rehabilitation in stroke (NeuroCog): study protocol for a randomized controlled trial. Trials. 2015 Sep 29;16:435. doi: 10.1186/s13063-015-0945-1. PMID 26420269